CLINICAL TRIAL: NCT02587507
Title: Proteomic Analysis of the Peripheral-Blood Mononuclear Cells Response After a High-Fat, High-Carbohydrate Meal With or Without Orange Juice in Healthy Subjects
Brief Title: Proteomic Analysis of Mononuclear Cells After a High-Fat, High-Carbohydrate Meal With or Without Orange Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Principal Investigator, Daniela Chaves, PhD, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TMTMNC
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Water; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Water (Placebo Comparator): The subjects will ingest the HFHC meal with 500mL of water.
  Interventions: Other: Water
- Orange juice (Experimental): The subjects will ingest the HFHC meal with 500mL of orange juice.
  Interventions: Other: Orange juice
- Water with glucose (Active Comparator): The subjects will ingest the HFHC meal with 500mL of water with glucose (isocaloric control of the orange juice).
  Interventions: Other: Water with glucose

INTERVENTIONS:
Other: Orange juice — Individuals will consume the HFHC meal with 500mL of orange juice.
  Arms: Orange juice
Other: Water — Individuals will consume the HFHC meal with 500mL of water.
  Arms: Water
Other: Water with glucose — Individuals will consume the HFHC meal with 500mL of water with glucose.
  Arms: Water with glucose

SUMMARY:
A high-fat, high-carbohydrate meal (HFHC) induces an increase in inflammation in peripheral-blood mononuclear cells in healthy subjects. A few studies have shown that orange juice, when consumed together with the high-fat meal, is able to revert the increase in inflammatory markers. The present study will assess the effect of a single HFHC meal taken with water, orange juice or an isocaloric glucose drink on protein expression in peripheral blood mononuclear cells of healthy individuals. Twelve healthy, normal weight individuals consumed a HFHC meal with water, water with glucose or orange juice in a cross-over design with at least one week interval between the meals. Blood samples were collected before, 1, 3 and 5h after the meals.

DETAILED DESCRIPTION:
BACKGROUND:

A high-fat, high-carbohydrate meal (HFHC) induces an increase in inflammation in peripheral-blood mononuclear cells in healthy subjects. A few studies have shown that orange juice, when consumed together with the high-fat meal, is able to revert the increase in inflammatory markers.

OBJECTIVES:

To study the effect of a single HFHC meal taken with water, orange juice (500ml) or an isocaloric glucose drink on protein expression in peripheral blood mononuclear cells of healthy individuals.

DESIGN AND METHODOLOGY:

Twelve healthy, normal weight individuals consumed a HFHC meal with water, water with glucose or orange juice in a cross-over design with at least one week interval between the meals. Blood samples were collected before, 1, 3 and 5h after the meals. Blood glucose, insulin and lipid profile were measured. Also, proteome analysis using TMT labeling was performed on peripheral-blood mononuclear cells collected before and at times 3 and 5h after the meal.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normal weight
* non-vegetarian

Exclusion Criteria:

* use of medication
* alcohol consumption,
* intense physical exercise
* pregnant or lactating
* overweight
* obese
* drug abuse
* any disease such as diabetes, inflammatory conditions.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in protein expression at mononuclear cells of healthy individuals before and after the high fat meal using TMT labeling and mass spectrometry | before the meal, 1h, 3h and 5h after the meal

SECONDARY OUTCOMES:
Blood glucose | before the meal
Blood glucose | 1h after the meal
Blood glucose | 3h after the meal
Blood glucose | 5h after the meal
Insulin | before the meal
Insulin | 1h after the meal
Insulin | 3h after the meal
Insulin | 5h after the meal
Lipid profile | before the meal
  total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides
Lipid profile | 1h after the meal
  total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides
Lipid profile | 3h after the meal
  total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides
Lipid profile | 5h after the meal
  total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Daniela FS Chaves, PhD, Principal Investigator — University of Sao Paulo

REFERENCES:
- [Result] Ghanim H, Sia CL, Upadhyay M, Korzeniewski K, Viswanathan P, Abuaysheh S, Mohanty P, Dandona P. Orange juice neutralizes the proinflammatory effect of a high-fat, high-carbohydrate meal and prevents endotoxin increase and Toll-like receptor expression. Am J Clin Nutr. 2010 Apr;91(4):940-9. doi: 10.3945/ajcn.2009.28584. Epub 2010 Mar 3. PMID 20200256
- [Result] Coelho RC, Hermsdorff HH, Bressan J. Anti-inflammatory properties of orange juice: possible favorable molecular and metabolic effects. Plant Foods Hum Nutr. 2013 Mar;68(1):1-10. doi: 10.1007/s11130-013-0343-3. PMID 23417730
- [Derived] Chaves DFS, Carvalho PC, Brasili E, Rogero MM, Hassimotto NA, Diedrich JK, Moresco JJ, Yates JR 3rd, Lajolo FM. Proteomic Analysis of Peripheral Blood Mononuclear Cells after a High-Fat, High-Carbohydrate Meal with Orange Juice. J Proteome Res. 2017 Nov 3;16(11):4086-4092. doi: 10.1021/acs.jproteome.7b00476. PMID 28927270